CLINICAL TRIAL: NCT05542459
Title: Multi-omics to Predict Responses to Biologics in Inflammatory Bowel Disease
Brief Title: Multi-omics to Predict Responses to Biologics in IBD
Acronym: MORE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Gao, Director, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2022ZSLYEC-136
Record Dates: First submitted 2022-09-10; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood, serum, white cells, urine, feces, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-IBD control group: A control group in which patients are not diagnosed as inflammatory bowel disease.
- CD group: A group in which patients are diagnosed as crohn's disease
  Interventions: Drug: Biologics
- UC group: A group in which patients are diagnosed as ulcerative colitis
  Interventions: Drug: Biologics

INTERVENTIONS:
Drug: Biologics — Infliximab, adalimumab, vedolizumab, ustekinumab, and other biologics approved for IBD
  Groups: CD group; UC group

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic immune-related disease, which mainly affects the digestive tract. There are mainly two forms of the disease, including Crohn's disease (CD) and ulcerative colitis (UC).

Biologics have revolutionized the treatment of inflammatory bowel disease with good efficacy and safety. However, 20-50% of patients may not response to or lose response to biologics. Unfortunately, there has been no factors or measures that may predict the efficacy or safety of biologics.

In this study, a large prospective cohort study is conducted to evaluate the efficacy and safety of biologics (infliximab, adalimumab, vedolizumab, ustekinumab, and other approved biologics) in patients with inflammatory bowel disease in the real clinical practice. Meanwhile, a multi-omics approach involving transcriptomics, microbiome, proteomics, and metabolome, are adopted to explore biomarkers or factors that predict the therapeutic efficacy or safety of biologics. The mechanism underlie the disease will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. For patients with IBD:

   * Patients with IBD treated with approved biologics
   * Age 18 or over
   * Written informed consent obtained from patient for participation
2. For non-IBD healthy volunteers:

   * Patients without the diagnosis of IBD or other conditions that, in the opinion of the investigator, not suitable to participate in the study
   * Age 18 or over
   * Written informed consent obtained from patient for participation

Exclusion Criteria:

* Unable to obtain written informed consent
* Patient is, in the opinion of the investigator, not suitable to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease treated with approved biologics
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response | At week 14-26
  The reduction of Crohn's Disease Activity Index (CDAI) ≥70 or CDAI <150 for Crohn's disease; a reduction of the Mayo Clinical Score ≥2 for ulcerative colitis
Mucosal healing | At week 42-64
  Mucosal healing is defined as absence of mucosal ulceration

SECONDARY OUTCOMES:
Clinical response rate with steroids or without steroids | At week 14-26 and week 42-64
  Clinical response rate with steroids or without steroids at week 14-26 and week 42-64
Clinical remission rate with steroids or without steroids | At week 14-26 and week 42-64
  Clinical remission rate with steroids or without steroids at week 14-26 and week 42-64
Objective response rate | At week 14-26 and week 42-64
  Objective response was defined based on results obtained from at least 1 among endoscopy, bowel ultrasound, and computerized tomography (CT) or magnetic resonance (MR) enteroclysis at week 14-26 and week 42-64
Objective remission rate | At week 14-26 and week 42-64
  Objective remission was defined based on results obtained from at least 1 among endoscopy, bowel ultrasound, and computerized tomography (CT) or magnetic resonance (MR) enteroclysis at week 14-26 and week 42-64
Inflammatory Bowel Disease Questionnaire (IBDQ) score | At baseline, week 14-26 and week 42-64
  IBDQ score at baseline, week 14-26 and week 42-64
36-Item Short Form Health Survey (SF-36) score | At baseline, week 14-26 and week 42-64
  SF-36 score at baseline, week 14-26 and week 42-64
EQ-5D score | At baseline, week 14-26 and week 42-64
  EQ-5D score at baseline, week 14-26 and week 42-64
Incidence of adverse events | Through study completion
  Incidence of adverse events through study completion

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li Q, Huang Z, Yang H, Tang J, Zuo T, Yang Q, Huang Z, Guo Q, Li M, Gao X, Chao K. Intestinal mRNA expression profiles associated with mucosal healing in ustekinumab-treated Crohn's disease patients: bioinformatics analysis and prospective cohort validation. J Transl Med. 2024 Jun 26;22(1):595. doi: 10.1186/s12967-024-05427-w. PMID 38926732